CLINICAL TRIAL: NCT05632770
Title: A Deployment Focused Pragmatic Trial of Optimal Stepped Care Intervention Targeting PTSD and Comorbidity for Acutely Hospitalized Injury Survivors Treated in US Trauma Care Systems
Acronym: TSOS 8
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, Psychiatry & Behavioral Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00015632; R01MH130460 (NIH)
Record Dates: First submitted 2022-11-17; First posted 2022-12-01 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: PTSD; Physical Injury
Keywords: PTSD; Physical Injury; Emergency Department Utilization
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Referral and Consultation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stepped Collaborative Care (Intervention) (Experimental): Patients in the intervention condition will receive a stepped collaborative care intervention that includes posttraumatic concern elicitation, proactive care management, medication, and psychotherapy elements targeting posttraumatic stress disorder (PTSD) and related comorbidity.
  Interventions: Behavioral: Stepped Collaborative Care
- American College of Surgeons (ACS) Required Screening and Referral (Usual Care) (Active Comparator): Patients in the control condition will receive usual trauma center care with American College of Surgeons (ACS) required psychosocial screening and referral.
  Interventions: Behavioral: American College of Surgeons (ACS) Required Screening and Referral (Usual Care)

INTERVENTIONS:
Behavioral: Stepped Collaborative Care — Case management, behavioral intervention elements, psychopharmacologic medication recommendations and 24/7 cell phone coverage for 6 months post-injury.
  Arms: Stepped Collaborative Care (Intervention)
Behavioral: American College of Surgeons (ACS) Required Screening and Referral (Usual Care) — The study will contribute to usual care with the study 10-domain electronic health record (EHR) screen and the posttraumatic stress disorder (PTSD) evaluation. The study team may also collaborate with hospital providers on the referral process and/or inform a member of the patient's care team of distress patients are experiencing as identified by a DSM-5 PTSD Checklist (PCL) score of ≥ 30 or a DSM-IV PTSD Checklist (PCL) score of ≥ 35.
  Arms: American College of Surgeons (ACS) Required Screening and Referral (Usual Care)

SUMMARY:
This investigation is a randomized pragmatic trial of a brief stepped care intervention delivered from an acute care medical trauma center that may both reduce the symptoms of posttraumatic stress disorder (PTSD) and diminish emergency department health service utilization.

DETAILED DESCRIPTION:
Life-threatening traumatic exposures requiring presentation to acute care medical settings are endemic in the US in the era of the COVID-19 pandemic, firearm proliferation, and extreme weather events, and constitute both a substantial source of individual suffering and a significant public health burden. Each year in the US, over 30 million individuals present to acute care medical settings after injury, and approximately 2.5 million individuals are so severely injured that they require inpatient hospital admissions. The overarching goal of the Trauma Survivors Outcomes and Support (TSOS) investigation is to advance the sustainable delivery of high quality trauma center mental health screening, intervention and referral procedures for diverse injury survivors. Over the past two decades, the TSOS study team that includes research scientists, trauma surgical policymakers, patients, and frontline clinicians has established a track record of using evidence derived from NIH pragmatic trials to directly target American College of Surgeons Committee on Trauma (College) regulatory policy. The TSOS investigation will refine and test optimal stepped care intervention strategies for diverse injury survivors presenting to acute care medical settings with PTSD and associated comorbidity. This single trauma center site pragmatic trial investigation will individually randomize 424 patients (212 intervention and 212 control) to a brief stepped care intervention versus College required screening and referral control conditions. The stepped care intervention consists of proactive care management, as well as medications and psychotherapy elements targeting PTSD and comorbidity. Blinded follow-up interviews at 1-, 3-, 6-, and 12-months post-injury will assess the symptoms of PTSD and related comorbidity for all patients. The emergency department health information exchange will be used to capture population-level automated emergency department/inpatient utilization data for the intent-to-treat sample. The investigation aims to test the primary hypotheses that intervention patients will demonstrate significant reductions in PTSD symptoms and emergency department/inpatient utilization when compared to control patients. The investigation will also explore mediators and moderators of intervention treatment effects that directly address actionable national trauma center quality improvements. A mixed method Rapid Assessment Procedure-Informed Clinical Ethnography (RAPICE) implementation process assessment will facilitate the integration of study results into national College policy requirements, guidelines, and verification criteria. A national trauma center survey will elucidate the progression of PTSD and comorbidity screening, intervention and referral for all US level I and II trauma centers. An end-of-study College policy summit will harness pragmatic trial data to inform the capacity for US trauma centers to implement high quality acute care medical mental health services for diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Injured patients ≥18 years of age
* Meet ≥ 3 of 10 risk domain criteria in electronic health records (EHR) screen
* Score of ≥ 30 on DSM-5 PTSD Checklist (PCL) score or score of ≥ 35 on DSM-IV PTSD Checklist (PCL) .
* Speak English and/or Spanish

Exclusion Criteria:

* Age <18
* Not admitted for a traumatic injury
* Speak a language other than English and/or Spanish
* Acutely suicidal/admitted for a suicide attempt
* Cognitively impaired
* Incarcerated
* Acutely psychotic
* Not a resident of Washington, California, Alaska, Oregon, Idaho, Montana, or Nevada
* Less than 2 pieces of contact information
* Prior history of violence, such that study staff may not be safe
* Patient with overwhelming psychiatric distress and not advisable/will not tolerate randomization to control condition
* Most recent COVID-19 test positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder (PTSD) symptoms change over time | Change in symptoms at baseline injury admission and 1-, 3-, 6-, and 12-months post-injury follow-up
  The investigators will use the DSM-5 PTSD Checklist (PCL-5) and DSM-IV PTSD Checklist (PCL-IV). The scoring of the PCL-5 scale ranges from a minimum of 0 to a maximum of 80, with higher scores indicating a worse outcome. The measure can also provide a rating of symptoms consistent with a diagnosis of PTSD.
Emergency department utilization change over time | Baseline injury admission to 12-months post-injury follow-up
  Number of emergency visits will be assessed using the Emergency Department Information Exchange (EDIE). More emergency visits are indicative of a worse outcome.

SECONDARY OUTCOMES:
Alcohol use change over time | Change in symptoms at baseline injury admission and 1-, 3-, 6-, and 12-months post-injury follow-up
  The investigators will use the Alcohol Use Disorders Identification Test - Concise (AUDIT-C) measure. The 3-item scale score ranges from 0-12, with higher values indicating a worse outcome.
Mental and physical functioning change over time | Change in symptoms at baseline injury admission and 1-, 3-, 6-, and 12-months post-injury follow-up
  The Medical Outcomes Study Short Form healthy survey (SF-12) will be used as a continuous measure. The 12-item scale score ranges from 0-100, with higher scores representing a better outcome. The two summary measures, Physical Component Summary (PCS) and Mental Component Summary (MCS), will be scored.
Depression symptoms change over time | Change in symptoms at baseline injury admission and 1-, 3-, 6-, and 12-months post-injury follow-up
  The Patient Health Questionnaire 9-item Depression Scale (PHQ-9) will be used to assess symptoms of depression. The scoring of the scale ranges from 0-27, with higher scores indicating a worse outcome. The scale can also be dichotomized to indicate depressive symptom cutoffs and DSM depressive disorder criteria.
Suicide risk assessment change over time | Change in symptoms at baseline injury admission and 1-, 3-, 6-, and 12-months post-injury follow-up
  The Columbia Suicide Severity Rating Scale (CSSRS) is a 6-item questionnaire to assess risk of suicide. The scoring of the scale ranges from 2-25, with higher scores indicating a worse outcome.
Substance use change over time | Change in symptoms at baseline injury admission and 1-, 3-, 6-, and 12-months post-injury follow-up
  Single items self report that assesses opioid use, amphetamines, cocaine and marijuana. Single item self-report are categorically rated from no use to use four or more times a week.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Knutzen T, Bulger E, Iles-Shih M, Hernandez A, Engstrom A, Whiteside L, Birk N, Abu K, Shoyer J, Conde C, Ryan P, Wang J, Russo J, Heagerty P, Palinkas L, Zatzick D. Stepped collaborative care versus American College of Surgeons Committee on Trauma required screening and referral for posttraumatic stress disorder: Clinical trial protocol. Contemp Clin Trials. 2024 Jan;136:107380. doi: 10.1016/j.cct.2023.107380. Epub 2023 Nov 10. PMID 37952714

DOCUMENTS (1):
  • Informed Consent Form (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/70/NCT05632770/ICF_000.pdf